CLINICAL TRIAL: NCT02276469
Title: Randomized Controlled Trial of Peer to Peer Support for People With Severe Mental Disorders: Schizophrenia, Affective Disorders and Personality Disorders in Comparison to Standard Care
Brief Title: Peer Support for Severe Mental Disorders
Acronym: PEER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Bock, Prof.Dr., Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC 0748/006; Psychenet Teilprojekt 5 (Other: University medicalcenter hamburg-eppendorf)
Record Dates: First submitted 2014-10-09; First posted 2014-10-28 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Psychosis; Major Depression; Bipolar Disorder; Borderline Personality Disorder
Keywords: severe mental illness
MeSH Terms: conditions — Psychotic Disorders; Depressive Disorder, Major; Bipolar Disorder; Borderline Personality Disorder; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- peer support (Experimental): peer support is delivered on individual basis for half a year, the frequency depends on the patients requirement, but at least 3 sessions has to occur
  Interventions: Behavioral: peer support
- usual care (No Intervention): usual care was delivered to the patients

INTERVENTIONS:
Behavioral: peer support — peer support is delivered by persons with a severe mental illness after the experience of recovery and after absolving a one year education to support others on their way to recovery
  Arms: peer support

SUMMARY:
The purpose of this study is to determine wether peer support is effective for the treatment of people with severe mental illness.

DETAILED DESCRIPTION:
A randomized controlled multi center trial is conducted, where patients receive usual care in the control group and usual care with additional peer support for 6 month in the intervention group. Psychosocial outcome criteria are collected pre intervention, after 6 month intervention and at one year follow up. Days till hospitalization and days spent in hospital are collected for one year before recruitment and one year after recruitment.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of schizophrenia, unipolar depression, bipolar disorder, personality disorder

Exclusion Criteria:

* primary clinical diagnosis of addiction

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-07; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Self-Efficacy at 6 month | 1. Baseline; 6 month follow up (post intervention); twelve month follow
  General Self-Efficacy Scale; Self report Questionnaire; 10 Items

SECONDARY OUTCOMES:
Change from Baseline in Quality of life at 6 and 12 month | 1. Baseline; 2. Six month follow up (post intervention) 3. Twelve month follow
  Self report questionnaires: Modulares System zur Lebensqualität MSLQ-R
Change from Baseline in Quality of life at 6 and 12 month | 1. Baseline; 2. Six month follow up (post intervention) 3. Twelve month follow
  Self report questionnaires: EuroQol-Group: EQ5D
Service satisfaction after six month of intervention | After six month intervention
  Self report questionnaire: Client Satisfaction Questionnaire CSQ 8
Change from Baseline in Illness management, Coping at 6 and 12 month | 1. Baseline; 2. Six month follow up (post intervention) 3. Twelve month follow
  FKV-LIS Freiburger Self report questionnaire: Fragebogen zur Krankheitsverarbeitung; examining coping strategies
Change from Baseline in Psychosocial functioning at 6 and 12 month | 1. Baseline; 2. Six month follow up (post intervention) 3. Twelve month follow
  Clinical observation: Global assessment of functioning DSM
Change from Baseline in Severity of illness at 6 and 12 month | 1. Baseline; 2. Six month follow up (post intervention) 3. Twelve month follow
  Clinical observation: Clinical global impression
Change from Baseline in Illness management, Coping at 6 and 12 month | 1. Baseline; 2. Six month follow up (post intervention) 3. Twelve month follow
  Self report questionnaire: Subjective sense of psychosis
Hospitalization in days of in-patient care | one year before, until one year past intervention
  The days of in patient care assessed from the clinical records
Days to hospitalization | Baseline until 12 month follow up
  Days to hospitalization after the beginning of treatment assessed from the clinical records

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bock, Prof. Dr., Principal Investigator — University Medical Center Hamburg-Eppendorf (UKE)

REFERENCES:
- [Background] Schwarzer, R., & Jerusalem, M. (1995). Generalized Self-Efficacy scale. In J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs (pp. 35- 37). Windsor, England: NFER-NELSON.
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Pukrop, R. (2003). Modulares System zur Lebensqualität. In J. Schumacher, A. Klaiberg & E. Brähler (Hrsg.), Diagnostische Verfahren zu Lebensqualität und Wohlbefinden (S. 227-232). Göttingen Bern Toronto S
- [Background] National Institute of Mental Health (1976). 028 CGI. Clinical Global Impressions. In: Guy, W. (Ed.), ECDEU Assessment for psychopharmacology. Rev. Ed. Rockville, Maryland. 217-222.
- [Background] Muthny FA. [References for evaluation scales in quality assurance in rehabilitation--6. Assessment of coping processes with the Freiburg Questionnaire of Illness Coping]. Rehabilitation (Stuttg). 1996 May;35(2):IX-XVI. German. PMID 8767546
- [Background] Sass, H., Wittchen, H.U., Zaudig, M. (2001). Diagnostisches und Statistisches Manual psychischer Störungen DSM-IV. Göttingen, Bern, Toronto, Seattle: Hogrefe Verlag für Psychologie
- [Background] Bock T, Brysinski T, Klapheck K, Bening U, Lenz A, Naber D. [On subjective meaning of psychoses. Construction, validation and first application of a new questionnaire--the SuSi-Project (Hamburg)]. Psychiatr Prax. 2010 Sep;37(6):285-91. doi: 10.1055/s-0030-1248424. Epub 2010 Jun 15. German. PMID 20552540